CLINICAL TRIAL: NCT01702285
Title: A Phase I Open Label, Multicenter, Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of Orally Administered CUDC-101 in Subjects With Advanced and Refractory Solid Tumors
Brief Title: Phase I Study to Assess the Safety, Tolerability, and Pharmacokinetics of Orally Administered CUDC-101 in Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUDC-101-105
Record Dates: First submitted 2012-09-25; First posted 2012-10-08 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Cancer
Keywords: Advanced Solid Tumors; EGFR; HDAC; Her2; Open-Label; Dose-Escalation
MeSH Terms: conditions — Neoplasms | interventions — 7-(4-(3-ethynylphenylamino)-7-methoxyquinazolin-6-yloxy)-N-hydroxyheptanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CUDC-101 (Experimental): 200-500 mg CUDC-101, orally administered, twice daily, in continuous 21 day cycles until disease progression or other discontinuation criteria are met.
  Interventions: Drug: CUDC-101

INTERVENTIONS:
Drug: CUDC-101 — 200-500 mg CUDC-101, orally administered, twice daily, in continuous 21 day cycles until disease progression or other discontinuation criteria are met.

SUMMARY:
The main purpose of this study is to determine the safety and tolerability of orally administered CUDC-101 in cancer patients, and to determine a dose for further testing. This study will also determine how well CUDC-101 is absorbed into the blood after being given orally, assess CUDC-101 blood levels and what happens to the study drug in the body, and study how the body reacts to the study drug and what effects it has on tumors. CUDC-101 has been administered to cancer patients as an intravenous (IV) infusion in other research studies, but has not been studied when given orally.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a histopathologically confirmed diagnosis of advanced solid tumor.
2. Subjects must have no further standard of care options.
3. Measurable or non-measurable disease
4. Age ≥ 18 years
5. ECOG performance status ≤ 2
6. Life expectancy ≥ 3 months
7. Women of child bearing potential must have a negative serum pregnancy test.
8. Absolute neutrophil count ≥ 1,500/µL; platelets ≥ 100,000/µL; creatinine ≤ 1.5x upper limit of normal (ULN); total bilirubin ≤ 1.5x ULN; AST/ALT ≤ 2.5x ULN. For subjects with documented liver metastases, the AST/ALT may be ≤ 5x ULN
9. Serum magnesium and potassium within normal limits (may be supplemented to achieve normal values).
10. Subjects with brain metastases are eligible if controlled on a stable dose of ≤ 10mg prednisone/day or its equivalent dose of steroids.
11. Men and women of child bearing potential must agree to use adequate birth control throughout their participation in the study and for 60 days following the last study treatment.
12. Able to provide written informed consent and to follow protocol requirements.

Exclusion Criteria:

1. Systemic anticancer therapy within 28 days prior to study treatment. Subjects with prostate cancer on LHRH hormonal therapy may be enrolled and continue on this therapy.
2. Use of any investigational agent(s) within 21 days prior to study treatment.
3. Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
4. Subjects receiving moderate or strong CYP3A4 or CYP2D6 inhibitors within 7 days prior to study treatment (See Appendix C for examples).
5. Serious infection requiring systemic antibiotic therapy within 14 days prior to study treatment.
6. Known gastrointestinal condition that would interfere with swallowing or the oral absorption or tolerance of CUDC-101.
7. Ongoing diarrhea of any grade (per NCI CTCAE v4.03).
8. Uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months prior to study treatment, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, or cardiac amyloidosis.
9. Unstable or clinically significant concurrent medical condition that would, in the opinion of the Investigator, jeopardize the safety of a subject and/or their compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and recommended Phase 2 dose of oral CUDC-101 in subjects with advanced and refractory solid tumors | 21 days (1 cycle of study treatment)
  The highest dose level studied at which fewer than 2 out of 6 subjects (< 33%) experience a dose limiting toxicity (DLT).
Assess the bioavailability (BA) of orally administered CUDC-101 | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours post-dose on the first and second day of study drug dosing.
  Comparison of area under the plasma concentration time curve (AUC) following intravenous and oral administrations.
Assess the pharmacokinetics (PK) of orally administered CUDC-101 | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours post-dose on the ninth day of study drug dosing
  Pharmacokinetic parameters will include AUC, maximum plasma concentration (Cmax),half-life (T1/2), clearance (Cl) and volume of distribution (Vd).

SECONDARY OUTCOMES:
Assess the safety and tolerability of continuous orally administered CUDC-101 | 18 months
  Number of participants with adverse events assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE, v4.0).
Evaluate biomarkers of CUDC-101 activity | Day 1 and Day 7 of Cycle 1 dosing.
  Pre- and post-dose changes in acetylated histone H3 protein levels in peripheral blood mononuclear cells (PBMCs), as well as skin and tumor biopsy samples (where available).
Assess preliminary anti-cancer activity | 18 months
  Occurrences of complete response, partial response, stable disease and progressive disease as determined by the Response Evaluation Criteria In Solid Tumors (RECIST v1.1).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Southern Texas Accelerated Research Therapeutics, San Antonio, Texas